CLINICAL TRIAL: NCT02171845
Title: Mechanisms and Factors Responsible for the Inhibition of Transposons During Fetal Gonad Development in Humans
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Other Study IDs: FAUQUE ANR 2011
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Medical Termination of Pregnancy; Voluntary Termination of Pregnancy
Keywords: Male foetuses of 10 to 37 weeks

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Foetus
  Interventions: Other: surgical biopsies

INTERVENTIONS:
Other: surgical biopsies

SUMMARY:
This is a single-centre study over 36 months for the inclusion of 30 patients. The selection and inclusion of patients will take place according to the criterion of Medical Termination of Pregnancy at 4 different gestational ages (8-12 weeks of gestation (WG)), 13-16 WG, 17-23 WG and 25-35 WG. The tissue analysed will principally be the gonads, other somatic tissue will also be systematically harvested in parallel (liver and psoas muscle) for control purposes. The gonads will be subjected to molecular biology analyses destined to quantify the expression of transposons and their inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Couple or mother who has provided written informed consent
* Foetus between 10 and 37 weeks of amenorrhea (WA)
* Male foetus
* Foetus obtained following medical termination of pregnancy or voluntary termination of pregnancy

Exclusion Criteria:

* persons without national health insurance cover
* foetus presenting aneuploidy
* foetus presenting a malformation of the genital organs

Ages: 10 Weeks to 37 Weeks | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Study Population: Male foetuses of 10 to 37 weeks of amenorrhea obtained following medical termination of pregnancy or voluntary termination of pregnancy.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-01-29 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Spatio-temporal analysis of the activity of TEs by RT-qPCR and immunostaining | Baselines

SECONDARY OUTCOMES:
Promoter methylation profile by pyrosequencing | Baselines

OTHER OUTCOMES:
Spatiotemporal analysis piARN way: RT qPCR, Small RNA Seq, and immunoprecipitation of proteins PIWI | Baselines

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de DIJON, Dijon, France